CLINICAL TRIAL: NCT03204110
Title: Non Invasive Assessment of Morphological and Functional Retinal Patterns in Reversible Cerebral Vasoconstriction Syndrome Using Transorbital Echotomography Doppler, Retinography and Retinal Vessel Analyser
Brief Title: Retinal Patterns in Reversible Cerebral Vasoconstriction Syndrome
Acronym: SVC-2R
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P100509
Record Dates: First submitted 2014-09-09; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Reversible Cerebrovascular Vasoconstriction Syndrome
Keywords: Reversible cerebral vasoconstriction syndrome; Anatomic and morphological retinal network analysis; Retinal vessel analyser; retinography; Prospective analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Reversible cerebral vasoconstriction syndrome (RCVS) is a clinico radiological entity characterized by severe headaches (associated or not with neurological complications) during one to 3 weeks, associated with a characteristic 'string and beads' appearance on cerebral arteries, which resolves spontaneously in 3 months. The pathway is unknown. At early stage of the disease (at the first medical consultation) cerebral arterial abnormalities which are necessary for diagnosis are identified in only 20% of patients (brain magnetic resonance imagery (MRI) ,CT scan angiography), appearing with a delay on 2th or 3rd week after the first severe headache..

Retinal artery network is considered to be a window on brain microvasculature by sharing the same embryologic origin and physiopathology. A retinal arteriolar examination at early stage of RCVS could provide non invasively early clue to confirm diagnosis by identifying anatomical change and /or functional abnormalities at the microvascular level, whereas large cerebral artery abnormalities are still normal.

DETAILED DESCRIPTION:
Reversible cerebral vasoconstriction syndrome (RCVS) is a clinico radiological entity characterized by severe headaches (associated or not with neurological complications) during one to 3 weeks, associated with a characteristic 'string and beads' appearance on cerebral arteries, which resolves spontaneously in 3 months.

The pathway is unknown. One strong hypothesis is that RCVS is a vasospasm and-vasodilatation disorder starting from small distal cerebral arteries progressing toward to medium sized and large sized cerebral arteries, and disappearing in 3 months.

At early stage of the disease (generally at the first medical consultation round 7 days after the first headache), arterial caliber anomalies cannot be identified on usual investigation (brain MRI, angioscan) in most of the case (80%). They are appearing secondary on repeated angiogram around the 2nd week or 3rd week, permitting to confirm the diagnosis, but with delay. Currently, small cerebral vessel arteries can't be studied directly . Retinal artery network is easy to study. It is considered to be a window on brain microvasculature by sharing the same embryologic origin and physiopathology. The investigators thus hypothesized that retinal arteriolar examination a early stage of RCVS could provide non invasively early clue to confirm diagnosis by identifying anatomical change and /or functional abnormalities at the microvascular level, whereas large cerebral artery abnormalities are still normal.

Hypothesis Arteriolar caliber and vasoreactivity abnormalities at the retinal microvascular level could be an early, non invasive and sensitive diagnostic marker of the RCVS at the first medical consultation in emergency.

ELIGIBILITY:
Inclusion Criteria:

* repetitive thunderclap headache highly suggestive of RCVS (clinical syndrome)
* maximum delay of ten days between the first thunderclap headache (qualifying event) and patient's inclusion.
* informed written consent

Exclusion Criteria:

* intracranial aneurism on angiography (Brain MRI or angioscan)
* severe atheroma with cervical stenosis up to 80%
* medical history of diabetes and/or hypertension
* minor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male and female with Reversible cerebral vasoconstriction syndrome
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-03-06 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2016-08-23 (Actual)

PRIMARY OUTCOMES:
The frequency of retinal morphological microvascular abnormalities | < 10 days
  The frequency of retinal abnormalities will be described at early stage of RCVS (< 10 days following the first thunderclap headache = qualifying event) • by measuring the retinal arteriolar caliber at baseline (micrometer, µm)
The frequency of retinal functional vascular abnormalities | < 10 days
  The frequency and type of retinal abnormalities will be described at early stage of RCVS (< 10 days following the first thunderclap headache = qualifying event) • by measuring the meanflow value in central retinal artery (cm/s), ciliar arteries (cm/s) and ophthalmic arteries(cm/s) at baseline
  • by measuring the diameter variation of retinal microvascular network (% of variation) during a vasoreactivity test (flicker stimulation with RVA)
The type of retinal morphological microvascular abnormalities | < 10 days
  The type of retinal abnormalities will be described at early stage of RCVS (< 10 days following the first thunderclap headache = qualifying event) • by measuring the retinal arteriolar caliber at baseline (micrometer, µm)
The type of retinal functional vascular abnormalities | < 10 days
  The type of retinal abnormalities will be described at early stage of RCVS (< 10 days following the first thunderclap headache = qualifying event) • by measuring the meanflow value in central retinal artery (cm/s), ciliar arteries (cm/s) and ophthalmic arteries(cm/s) at baseline
  • by measuring the diameter variation of retinal microvascular network (% of variation) during a vasoreactivity test (flicker stimulation with RVA)

SECONDARY OUTCOMES:
The kinetic of morphological retinal abnormalities during RCVS | at Day10, Day14, Day21 and Day 90
  The kinetic of morphological retinal abnormalities during RCVS course from the first neurological evaluation to final neurological follow up at 3 months (Day10, Day14, Day21 and Day 90) using the same morphological and functional measurements at the retinal level (RVA, retinography, and transorbital echo Doppler)
the kinetic of morphological patterns on Brain RMI during RCVS course during RCVS course | at Day10, Day 14, Day 21 and Day 90
  The kinetic of morphological patterns at the cerebral level: Brain RMI (Magnetic resonance Imaging) at Day10 Day14 Day21 and Day 90 : existence or not and number of vasopasm , existence or not of ischemic lesions, existence or not of hemorrhagic lesions.
the kinetic of functional patterns on cervico transcranial duplex evaluation during RCVS course | at Day10, Day 14, Day 21 and Day 90
  The kinetics of functional patterns at the cerebral level (men velocities cm/s for MCA CAA, BA, maximum systolic peak values on MCA, CAA and BA )using cervico transcranial duplex

CONTACTS AND LOCATIONS:
Overall Officials: GOBRON Claire, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Physiological department, Lariboisière hospital, Paris, France